CLINICAL TRIAL: NCT00968786
Title: A Trial of the Use of Multiple Automated Measuring Devices in the Management of Patients With Hypertension and Type 2 Diabetes Mellitus
Brief Title: Home Monitoring in the Management of Hypertension and Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Shanghai Institute of Hypertension, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HTDM 01
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2009-08-31 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
Keywords: hypertension; type 2 diabetes; home monitoring
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- no home monitoring (No Intervention): no automated measuring devices for patients use at home
  Interventions: Device: Home monitoring

INTERVENTIONS:
Device: Home monitoring — automated measuring devices for patients using at home

SUMMARY:
The home monitoring of automated measuring devices may improve the management of the chronic diseases, and may decrease the incidence of fatal disease. The investigators conducted a small sample and short observation time research to explore the feasibility to carry out later large-scale research.

DETAILED DESCRIPTION:
Background:

Approximately 40% of type 2 diabetes patients are also with hypertension. There are many risk factors in these patients, and so it's difficult to manage these patients. With the improvement of the accuracy of automated measuring devices, the patients can use these devices to monitor blood pressure, blood glucose, body weight, visceral fat and other indicators at home, and contribute their own participation in the management of there own diseases. The home monitoring may improve the management of this chronic disease, and may decrease the incidence of fatal disease such as stroke, myocardial infarction, heart failure, renal dysfunction and other serious diseases.

Large-scale research will carry out to prove that whether home monitoring is valuable for preventing the incidence of fatal disease such as stroke, myocardial infarction, heart failure, renal dysfunction. And in the first, it is necessary to conduct a small sample (n = 100), short observation time (six months) research, to monitor blood pressure, blood glucose, body weight and other indicators of intermediate target detection, to explore the feasibility to carry out such large-scale research.

Objective:

In hypertensive and type 2 diabetes patients, conducted an open randomized controlled trial to explore the patient's own use blood pressure monitors, blood glucose meter and pedometer at home, and use the body composition measurement instruments in clinic, is to be more effective control of blood pressure, blood glucose, body weight, and reduce the risk of patients with albuminuria.

Inclusion criteria:

1. Regardless of whether they are currently receiving antihypertensive therapy, systolic blood pressure higher than 140 mmHg or diastolic blood pressure higher than90 mmHg.
2. Whether or not use oral hypoglycemic agents or insulin injections, the fasting plasma is higher than 7.0 mmol/L, or postprandial blood glucose higher than 11.1 mmol/L.

Exclusion criteria:

1. with life-threatening disease.
2. With the various effects of metabolic diseases such as hyperthyroidism, hypothyroidism, etc.
3. stroke, myocardial infarction and other serious cardiovascular and cerebrovascular diseases occurred within 3 months.
4. serum creatinine level hugher than 176.8 mol/L.
5. Dementia or severe cognitive decline.
6. unable to do a long-term follow-up study or do not agree to participate in this trial.

Sample estimates and statistical analysis:

In accordance with 6-month follow-up, the average difference between the two groups, systolic blood pressure 3 mmHg, glycated hemoglobin 0.2%, under the conditions of a= 0.05 and b= 0.10, the research needs of each group of about 50 patients, a total of 100.

Major findings of the statistics using t test comparing the two groups after 6 months follow-up observations from the baseline change in the margin, and calculated 95% confidence interval. At the same time will also use non-parametric Wilcoxon test were compared blood pressure, blood glucose and so many follow-up results of repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

* Regardless of whether they are currently receiving antihypertensive therapy, systolic blood pressure higher than 140 mmHg or diastolic blood pressure higher than 90 mmHg.
* Whether or not use oral hypoglycemic agents or insulin injections, the fasting plasma is higher than 7.0 mmol/L, or postprandial blood glucose higher than 11.1 mmol/L.

Exclusion Criteria:

* With life-threatening disease.
* With the various effects of metabolic diseases such as hyperthyroidism, hypothyroidism, etc.
* Stroke, myocardial infarction and other serious cardiovascular and cerebrovascular diseases occurred within 3 months.
* Serum creatinine level higher than 176.8 mmol/L
* Dementia or severe cognitive decline
* Unable to do a long-term follow-up or do not agree to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
blood pressure, blood glucose, body weight and visceral fat levels. | 3,6 months

SECONDARY OUTCOMES:
albuminuria | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, Doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine